CLINICAL TRIAL: NCT07213115
Title: Epidemiology and Treatment of Gastric Cancer in the Federal State of Brandenburg From 2000 to 2020. An Analysis Using Data From the Clinical Cancer Registry for Brandenburg and Berlin.
Brief Title: Epidemiology and Treatment of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Collaborators: Margarete-Ammon-Stiftung (Unknown)
Responsible Party: Principal Investigator, Ulrike Weber, MSc., Medizinische Hochschule Brandenburg Theodor Fontane
Other Study IDs: EpiGaCa
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Gastric (Stomach) Cancer; Sex Difference
Keywords: Gastric Cancer; sex difference; registry data; epidemiology; treatment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sex
  Interventions: Procedure: Gastrectomy+ chemotherapy

INTERVENTIONS:
Procedure: Gastrectomy+ chemotherapy

SUMMARY:
According to recent statistics, the incidence and mortality from gastric cancer are both worldwide in fifth place in terms of ranking. Gastric cancer is more common in males than in females. This difference in the incidence between males and females is likely due to the difference in exposure to some risk factors like Helicobacter pylori infection, family history of gastric cancer, dietary habits, smoking and alcohol. However these factors do not completely explain the different characteristics of gastric cancer between the sexes. Some studies have concluded that exposure to estrogen could reduce the risk of gastric cancer.

There is a lack of current population based and real world data on sex and age differences in gastric cancer care. Analyses of sex differences are primarily originate from Asia or focusing on older cohorts. In the Netherlands, Kalff et al. conducted a study with patients with gastric adenocarcinoma (n=2 072) registered in the Dutch Upper GI Cancer Audit between 2011 and 2016. In this study, patients without metastatic gastric cancer and with an elective surgery were included.

To close this sex and age data gap for patients including those with UICC IV stage and without surgery, the aim of our study was to analyze the sex and age differences in clinicopathological features and staging in gastric adenocarcinoma with cancer registry data from the Federal State of Brandenburg from 2000 to 2020.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinomas (ICD-10-GM: C16.0 -C16.9)

Exclusion Criteria:

* missing age or sex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis focused on patients diagnosed with gastric adenocarcinomas (ICD-10-GM: C16.0 -C16.9) between 2000 and 2020 and residing in the Federal State Brandenburg. The data status was 31. December 2020. In the period between 2000 and 2020, a total of 8 582 patients residing in the state Brandenburg with newly diagnosed gastric adenocarcinoma were documented in the Cancer Registry and provided for the analysis in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8582 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 year, 10 year
  Survival time after date of cancer diagnosis

OTHER OUTCOMES:
sex differences | 5 year, 10 year
  Sex differences in epidemiology, Clinicopathological Characteristics, treatment, survival

IPD SHARING:
Plan to Share IPD: No